CLINICAL TRIAL: NCT02966275
Title: Closed-Loop Glucagon Administration For The Automated Treatment Of Post-Bariatric Hypoglycemia
Brief Title: Post Bariatric Closed Loop Glucagon Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P000710
Record Dates: First submitted 2016-05-10; First posted 2016-11-17 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Hypoglycemia
Keywords: glucagon; continuous glucose monitorering (CGM); artificial pancreas; hypoglycemia; post-bariatric hypoglycemia; bionic pancreas; bariatric surgery
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Glucagon and placebo were blinded by the research pharmacy. Subjects were given bags of blinded medication labeled with which day they were to be used, and then were asked to label the bags with which day the medication was actually used. The contents of the bags were verified with the research pharmacy's blinding key upon completion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Glucagon-only bionic pancreas - glucagon (Experimental): Subjects will wear the bionic pancreas that consists of a continuous glucose monitor linked to a smartphone running a hypoglycemia prevention algorithm that doses glucagon from an insulin pump through a subcutaneous infusion set.
  Subjects will continue to manage any hypoglycemia that occurs according to the current recommendations of their care provider.
  Interventions: Device: Glucagon-only bionic pancreas - glucagon
- Glucagon-only bionic pancreas - placebo (Placebo Comparator): Subjects will wear the bionic pancreas that consists of a continuous glucose monitor linked to a smartphone running a hypoglycemia prevention algorithm that doses placebo from an insulin pump through a subcutaneous infusion set.
  Subjects will continue to manage any hypoglycemia that occurs according to the current recommendations of their care provider.
  Interventions: Device: Glucagon-only bionic pancreas - placebo

INTERVENTIONS:
Device: Glucagon-only bionic pancreas - glucagon — A computer algorithm will automatically deliver glucagon based on the signal from a minimally invasive continuous glucose monitor.
  Arms: Glucagon-only bionic pancreas - glucagon
Device: Glucagon-only bionic pancreas - placebo — A computer algorithm will automatically deliver placebo based on the signal from a minimally invasive continuous glucose monitor.
  Arms: Glucagon-only bionic pancreas - placebo

SUMMARY:
This study is to test our automated hypoglycemia prevention and treatment device (glucagon-only bionic pancreas) in subjects that have undergone post-bariatric surgery that are experiencing symptoms of hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years or older with a gastric bypass for more than 1 year.
* Post-bariatric hypoglycemia with prior episodes of neuroglycopenia, unresponsive to dietary intervention (low glycemic index, controlled carbohydrate portions) and trial of acarbose therapy at the maximally tolerated dose. Other therapies will not exclude a subject as long as the therapy is continued during the study.
* Otherwise healthy (mild chronic disease such as asthma, hypertension, and depression will be allowed if well controlled).
* Self-reported frequency of documented hypoglycemia (BG < 60 mg/dl verified by capillary blood glucose measurements) of at least 2 times per week.

Exclusion Criteria:

* Unable to provide informed consent.
* Unable to comply with study procedures.
* Current participation in another hypoglycemia related clinical trial other than one that is primarily observational in nature.
* Pregnancy (positive urine HCG), breast feeding, plan to become pregnant in the immediate future, or sexually active without use of contraception.
* Use of insulin and/or insulin secretogues as sulfonylurea, metglitides, and glitazones.
* History of cystic fibrosis, pancreatitis, type 1 diabetes or other pancreatic disease.
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
* Any known liver or biliary disease including cirrhosis, alcoholic liver disease, non-alcoholic fatty liver disease, non-alcoholic steatohepatitis, any form of viral hepatitis.
* Congestive heart failure (established history of CHF, paroxysmal nocturnal dyspnea, or orthopnea).
* Acute illness or exacerbation of chronic illness at the time of the study.
* Known insulinoma or predominantly fasting pattern of hypoglycemia
* Adrenal insufficiency. Congenital hyperinsulinemia presenting with hypoglycemia during infancy.
* History of pheochromocytoma. Fractionated metanephrines will be tested in patients with history increasing the risk for a catecholamine secreting tumor:
* Paroxysms of tachycardia, pallor, or headache.
* Personal or family history of MEN 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease.
* Episodic or treatment refractory (requiring 4 or more medications to achieve normotension) hypertension.
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and/or any psychiatric hospitalization in the last year).
* Current alcohol abuse (intake averaging > 3 drinks daily in last 30 days) or substance abuse (any use within the last 6 months of controlled substances without a prescription).
* Unwilling or unable to refrain from drinking more than two drinks in an hour or more than four drinks in a day during the trial.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to RF interference.
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Unwilling or unable to completely avoid acetaminophen during the study period.
* Any factors that, in the opinion of the principal investigator, would interfere with the safe completion of the study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD, PhD, Principal Investigator — Massachusetts General Hospital, Boston, Massachusetts
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Information about this and related studies — http://bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 participants were enrolled in the trial and participated in the study
Groups:
- Glucagon-only Bionic Pancreas: Subjects will use the device every day and will fill the reservoir daily with glucagon or placebo (randomized, double blinded allocation for each day). Participants would be on glucagon or placebo for either 1 day or 2 days and then switch to the alternate arm. They could not be on the same arm for more than 2 days in a row.
  Glucagon-only Bionic Pancreas: A computer algorithm will automatically deliver glucagon based on the signal from a minimally invasive continuous glucose monitor.
Period: Overall Study
Arm/Group | Glucagon-only Bionic Pancreas
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All 10 participants who were enrolled in the study and completed the 14 day study period
Groups:
- Glucagon-only Bionic Pancreas: Subjects will use the device every day and will fill the reservoir daily with either glucagon or placebo (randomized, double blinded allocation for each day) for 14 days.
  Glucagon-only Bionic Pancreas: A computer algorithm will automatically deliver glucagon or placebo based on the signal from a minimally invasive continuous glucose monitor.
Arm/Group | Glucagon-only Bionic Pancreas
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Area Over the Curve and <60 mg/dl (CGM) Measured in mg/dl *Min
Description: The measure for area over the curve is used when an integrated assessment (e.g., a measurement of something over a specific amount of time) is more useful in understanding a phenomenon. To calculate this measure, a method of approximation is often used. One way would be to estimate the curve via curve-fitting techniques. For this outcome, using area over the curve and <60mg/dl provides a more robust method of calculating amount of hypoglycemia (by including more severe degrees of hypoglycemia in the product of mg/dl*min as opposed to percentage of time below 60mg/dl.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: mg/dl *minute
Groups:
- Glucagon-only Bionic Pancreas - Glucagon: Subjects will wear the bionic pancreas that consists of a continuous glucose monitor linked to a smartphone running a hypoglycemia prevention algorithm that doses glucagon from an insulin pump through a subcutaneous infusion set.
  Subjects will continue to manage any hypoglycemia that occurs according to the current recommendations of their care provider.
  Glucagon-only bionic pancreas - glucagon: A computer algorithm will automatically deliver glucagon based on the signal from a minimally invasive continuous glucose monitor.
- Glucagon-only Bionic Pancreas - Placebo: Subjects will wear the bionic pancreas that consists of a continuous glucose monitor linked to a smartphone running a hypoglycemia prevention algorithm that doses placebo from an insulin pump through a subcutaneous infusion set.
  Subjects will continue to manage any hypoglycemia that occurs according to the current recommendations of their care provider.
  Glucagon-only bionic pancreas - placebo: A computer algorithm will automatically deliver placebo based on the signal from a minimally invasive continuous glucose monitor.
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
mg/dl *minute | 1066.30 (2100.17) | 2004.80 (3076.93)

2. Secondary Outcome: Mean Continuous Glucose Monitor (CGM) Glucose
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
mg/dl | 112.3 (10) | 110.2 (11.74)

3. Secondary Outcome: Percentage of Time With CGM Glucose Less Than 60 mg/dl Overnight (11:00 PM - 7:00 AM)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 0.93 (1.41) | 3.95 (5.5)

4. Secondary Outcome: Percentage of Time With CGM Glucose Less Than 60 mg/dl During Daytime ( 7:00 AM-11:00 PM)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 1.43 (2.40) | 1.47 (1.85)

5. Secondary Outcome: Percentage of Time Spent Within the Glucose Range 70-120 mg/dl
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 66.53 (13.15) | 63.41 (15.00)

6. Secondary Outcome: Percentage of Time Spent Within the Glucose Range 70-180 mg/dl
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 92.67 (7.07) | 89.31 (8.22)

7. Secondary Outcome: Percentage of Time Spent Within the Glucose Range >180 mg/dl
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 4.27 (4.48) | 4.81 (4.41)

8. Secondary Outcome: Fraction of Time Spent Within the Glucose Range >250 mg/dl
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of time | 0.35 (0.66) | 0.10 (0.16)

9. Secondary Outcome: Mean Absolute Relative Deviation (MARD) of CGM vs. All StatStrip Xpress BG Measurements
Description: MARD is computed using the difference between the CGM readings and the values measured at the same time by the reference measurement system. The mean (or average) of all the absolute relative deviations produces the MARD. In this study, the reference measurement system was the StatStrip Xpress meter, to which the CGM values were compared.
Time Frame: 14 days
Population: The 2 arms are combined for this analysis as subjects switched arms either daily or every other day through the 14 days. During this period, subjects wore 2 sensors in total (1 sensor lasts 7 days). We do not expect a difference in accuracy resulting from switching arms this frequently or relating to glucagon vs placebo.
Measure: Mean (Standard Deviation); unit: percent difference
Groups:
- All Randomized Participants: All participants that were randomized and began participation in the trial
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 10
percent difference | 14.2 (12.5)

10. Secondary Outcome: Number of Carbohydrate Interventions for Hypoglycemia Per Day
Description: Number of carbohydrate interventions for hypoglycemia per day calculated from daily email survey
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: interventions/day
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
interventions/day | 1.17 (1.25) | 1.32 (0.94)

11. Secondary Outcome: Total Number of Grams of Carbohydrate Taken for Hypoglycemia Per Day
Description: Calculated from daily email survey
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
grams | 24.09 (26.10) | 22.56 (22.07)

12. Secondary Outcome: Total Glucagon Dosing (mcg/kg/24 Hours)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: mcg/kg/day
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
mcg/kg/day | 8.34 (3.76) | 10.1 (4.3)

13. Secondary Outcome: Number of Symptomatic Hypoglycemia Events Per Day
Description: Number of symptomatic hypoglycemia events per day calculated from daily email survey
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: events per day
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
events per day | 1.37 (1.05) | 1.56 (0.94)

14. Secondary Outcome: Percentage of Days When Participants Correctly Guessed Intervention (Glucagon vs Placebo) Out of a Total of 14 Days.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
percentage of days | 1.9 (1.5) | 1.4 (1.1)

15. Secondary Outcome: Number of Days With Nausea
Description: Number of days with nausea calculated from daily survey
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
days | 1.1 (1.6) | 1.1 (2.0)

16. Secondary Outcome: Severity of Nausea on Daily E-mail Survey
Description: The visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. We used a simple VAS is a straight horizontal line of fixed length measuring 0-100mm with subscale markings every 10mm. The ends are defined as the extreme limits of the parameter to be measured (nausea) orientated from the left (least severity or 0) to the right (most severity or 100mm). Subjects can mark their response anywhere from 0 to 100mm. The mean severity of nausea for the group in each arm was calculated by averaging all responses in either arm.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
Number analyzed (Participants) | 10 | 10
millimeters | 0.5 (0.7) | 0.5 (0.7)

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | Glucagon-only Bionic Pancreas - Glucagon | Glucagon-only Bionic Pancreas - Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/75/NCT02966275/Prot_SAP_000.pdf